CLINICAL TRIAL: NCT01082081
Title: A Study to Compare the Analgesic Efficacy of Two Different Paracetamol Doses as Measured by Post-operative Dental Pain Relief
Brief Title: Post-operative Dental Pain Study Comparing Analgesic Efficacy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4000684
Record Dates: First submitted 2010-02-18; First posted 2010-03-08 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-03

CONDITIONS: Post-surgical Dental Pain
Keywords: paracetamol; dental pain; Post-surgical dental pain
MeSH Terms: conditions — Toothache | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paracetamol 1000 mg (Experimental): Paracetamol 1000 mg
  Interventions: Drug: Paracetamol 1000 mg
- Paracetamol 500 mg (Experimental): Paracetamol 500 mg
  Interventions: Drug: Paracetamol 500 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol 1000 mg — Paracetamol 1000 mg
  Arms: Paracetamol 1000 mg
Drug: Paracetamol 500 mg — Paracetamol 500 mg
  Arms: Paracetamol 500 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
GlaxoSmithKline will be conducting this trial to compare analgesics efficacy of paracetamol 1000mg vs 500mg . The post-surgical dental pain model will be used to evaluate the analgesic efficacy of paracetamol. Each subject will be enrolled in the study for up to six weeks. The duration of the entire study will be approximately 16 weeks. Each subject will have to come to the clinic for three visits (Screening, Treatment and Follow up visits).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-45 years with moderate-to-severe dental pain assessed by verbal rating scale (VRS) and confirmed by a score of at least 50 mm out of 100 mm using a visual analogue scale (VAS) following surgical removal of third molars, of which at least one has to be a mandibular partially bony or full bony impaction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - PPD Dental Clinic, Austin, Texas
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Yue Y, Collaku A, Brown J, Buchanan WL, Reed K, Cooper SA, Otto J. Efficacy and speed of onset of pain relief of fast-dissolving paracetamol on postsurgical dental pain: two randomized, single-dose, double-blind, placebo-controlled clinical studies. Clin Ther. 2013 Sep;35(9):1306-20. doi: 10.1016/j.clinthera.2013.07.422. Epub 2013 Aug 22. PMID 23972577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Of 438 screened participants, 138 were considered to be screen failures. Remaining 300 were randomized to study treatments.
Groups:
- Paracetamol Caplet 1000 Milligrams (mg): Participants were administered with two paracetamol fast dissolving (FD) 500 mg caplets (total dose= 1000 mg), with 150 milliliter (mL) of water through oral route.
- Paracetamol Caplet 500 mg: Participants were administered with one paracetamol FD 500 mg caplet and one placebo caplet, with 150 mL of water through oral route.
- Placebo Caplet: Participants were administered with two placebo caplets, with 150 mL of water through oral route.
Period: Overall Study
Arm/Group | Paracetamol Caplet 1000 Milligrams (mg) | Paracetamol Caplet 500 mg | Placebo Caplet
Started | 121 | 119 | 60
Completed | 121 | 118 | 58
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other Reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracetamol Caplet 1000 mg: Participants were administered with two paracetamol FD 500 mg caplets (total dose= 1000 mg), with 150 mL of water through oral route.
- Total: Total of all reporting groups
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet | Total
Number analyzed (Participants) | 121 | 119 | 60 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.0 (5.0) | 23.9 (3.9) | 23.5 (4.9) | 23.9 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 73 | 37 | 178
  Male | 53 | 46 | 23 | 122
Number of participants with pain severity score measured on a rating scale [Number; unit: Participants] — Pain severity score was assessed on a 4-point categorical verbal rating scale. Total possible pain severity score range was none, mild, moderate and severe.
  Participants
    Moderate | 97 | 97 | 48 | 242
    Severe | 24 | 22 | 12 | 58

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Relief and Pain Intensity Differences From 0 to 6 Hours (SPRID 6 Hours)
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -5.8 (least pain relief) to 40.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief]
Time Frame: Every two hours from baseline to 6 hours post dose
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 10.60 (11.75) | 5.87 (9.03) | 3.35 (9.67)
Statistical Analysis 1: Comparison: Paracetamol Caplet 1000 mg vs Paracetamol Caplet 500 mg; Null hypothesis considered no difference in SPRID^6h between Paracetamol 1000 mg caplet and Paracetamol 500 mg caplet; Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA model included factors for treatment as a fixed effect and baseline assessment of pain intensity (VAS score) as a covariate; Adjusted Mean Difference = 4.77, 95% CI 2-sided [2.15 to 7.39] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: Paracetamol Caplet 1000 mg vs Placebo Caplet; Null hypothesis considered no difference in SPRID^6h between Paracetamol 1000 mg caplet and placebo caplet; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = 7.25, 95% CI 2-sided [4.04 to 10.45] — Difference was first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 3: Comparison: Paracetamol Caplet 500 mg vs Placebo Caplet; Null hypothesis considered no difference in SPRID^6h between Paracetamol 500 mg caplet and placebo caplet; Test type: Superiority or Other; p = 0.1307, ANCOVA; [statistical method as in outcome 1, analysis 1]; Adjusted Mean Difference = 2.48, 95% CI 2-sided [-0.74 to 5.69] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Time to Confirmed First Perceptible Pain Relief
Description: Participants recorded the time to first perceptible relief by starting the first stopwatch at the time of dosing and stopping it when he/she experienced the first perceptible pain relief. The first perceptible pain relief was confirmed if the participant also stopped the second stopwatch indicating meaningful relief.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received one study treatment and have at least one post-baseline efficacy assessment. Participants who did not achieve first perceptible pain relief during the 6 hours of the study period or took rescue medication were censored at the time 360 minutes.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
minutes | 80.63 (132.65) | 119.10 (156.44) | 189.53 (172.28)

3. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch when they first began to experience meaningful relief.
Time Frame: Baseline to 6 hours post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
minutes | 96.44 (128.64) | 129.75 (150.38) | 207.67 (162.01)

4. Secondary Outcome: Time to Start Using Rescue Medication
Description: Median time of use of rescue medication by participants was calculated.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received one study treatment and had at least one post-baseline efficacy assessment. Participants who did not achieve first perceptible pain relief during the 6 hours of the study period or took rescue medication were censored.
Measure: Median (Full Range); unit: minutes
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
minutes | 242.00 [92.00 to 360.00] | 189.00 [65.00 to 360.00] | 148.00 [61.00 to 360.00]

5. Secondary Outcome: Percentage of Participants Who Took Rescue Medication Within 2 Hours
Description: Percentage of participants who received rescue medication within 2 hours
Time Frame: Baseline to 2 hours post dose
Population: ITT population: All participants who received one study treatment and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Percentage of participants | 5.00 | 11.80 | 18.30

6. Secondary Outcome: Percentage of Participants Who Took Rescue Medication During 2 to 6 Hours
Description: Percentage of participants who took rescue medication during 2 to 6 hours
Time Frame: Within 2 to 6 hours post dose
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Percentage of participants | 57.9 | 55.5 | 53.3

7. Secondary Outcome: SPRID at 2 Hours
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -1.8 (least pain relief) to 12.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief]
Time Frame: Every two hours from baseline to 2 hours post dose
Population: ITT population: All participants who received study treatment and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 4.62 (3.31) | 3.26 (2.98) | 1.49 (2.54)

8. Secondary Outcome: SPRID at 4 Hours
Description: SPRID:Sum of Pain Intensity Difference (SPID) and Total Pain Relief (TOTPAR) at each post-dosing time-point. SPRID score ranged from -3.8 (least pain relief) to 26.3 (highest pain relief). SPID and TOTPAR were calculated as weighted sums of Pain Intensity Differences (PID) and Pain Relief Scores (PRS) at each measurement time, respectively. PID was derived by subtracting the pain severity score at a given post-dosing time-point from the baseline [pain severity score range:0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain using a 4-point categorical Verbal Rating Scale (VRS)]. If the subject rated pain intensity as 2 or 3, pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from baseline pain scores. PRS was assessed on 5-point categorical pain relief rating scale [0-no relief, 1-little relief, 2-some relief, 3-a lot of relief, 4-complete relief]
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 7.82 (7.36) | 4.42 (5.55) | 2.07 (5.45)

9. Secondary Outcome: Total Pain Relief (TOTPAR) at 2 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 2 hours post dose
Population: ITT population: All participants who received study treatment and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 3.33 (1.98) | 2.46 (1.81) | 1.47 (1.53)

10. Secondary Outcome: TOTPAR at 4 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 5.82 (4.37) | 3.73 (3.32) | 2.55 (3.15)

11. Secondary Outcome: TOTPAR at 6 Hours
Description: TOTPAR was calculated as sum of products of pain relief (PR) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240, 240-300 and 300-360. Higher score indicated greater pain relief.
  TOTPARt = ∑PR x (timet - timet-1).
  PR score was assessed at each of the above time-points based on a 5-point categorical scale [0-no relief, 1-little relief, 2-meaningful relief, 3-a lot of relief, 4-complete relief].
Time Frame: Every two hours from baseline to 6 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 8.05 (7.00) | 5.18 (5.44) | 4.10 (5.72)

12. Secondary Outcome: Sum of Pain Intensity Difference (SPID) Scores at 2 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 2 hours post dose
Population: ITT population: All participants who received study treatment and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 1.3 (1.5) | 0.8 (1.3) | 0.0 (1.2)

13. Secondary Outcome: SPID Scores at 4 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 4 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 2.0 (3.3) | 0.7 (2.6) | -0.5 (2.6)

14. Secondary Outcome: SPID Scores at 6 Hours
Description: SPID was calculated as sum of products of Pain Intensity Differences (PID) at a given time-point (t) with the time-interval from that time-point to the previous time-point (t-1). The time-intervals used were 0-15, 15-30, 30-45, 45-60, 60-90, 90-120, 120-240, 240-300 and 300-360. Positive and higher scores indicate greater reduction in pain.
  SPIDt = ∑PID x (timet - timet-1)
  Pain Intensity was assessed at baseline and at each time-point based on a 4-point categorical Verbal Rating Scale (VRS) scale: 0-no pain, 1-mild pain, 2-moderate pain, 3-severe pain.
  If the subject rated pain intensity as "2" or "3", pain was assessed using a 100 mm Visual Analog Scale (VAS) [0 (no pain), 100 (worst pain)]. VAS scores were converted into PID scores by subtracting them from pain scores taken at baseline.
Time Frame: Every two hours from baseline to 6 hours post dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 2.6 (5.1) | 0.7 (4.1) | -0.8 (4.4)

15. Secondary Outcome: Participants Global Assessment to Response to Treatment (PGART)
Description: PGART was measured by a score in a scale from 0-4: 0- Poor; 1- Fair 2- Good; 3- Very Good; 4- Excellent.
Time Frame: Baseline to 6 hours post dose
Population: ITT population: All participants who received study treatment and had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Number analyzed (Participants) | 121 | 119 | 60
Units on a scale | 1.54 (1.20) | 1.24 (1.11) | 0.63 (0.92)

ADVERSE EVENTS:
Time Frame: All adverse events encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | Paracetamol Caplet 1000 mg | Paracetamol Caplet 500 mg | Placebo Caplet
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/119 | 0/60
Other Adverse Events (participants affected / at risk) | 32/121 | 25/119 | 9/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracetamol Caplet 1000 mg (N=121) | Paracetamol Caplet 500 mg (N=119) | Placebo Caplet (N=60)
Alveolar Osteitis (Infections and infestations) | 20 (20) | 18 (18) | 3 (3)
Headache (Nervous system disorders) | 12 (13) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.